CLINICAL TRIAL: NCT07158996
Title: An Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Preliminary Clinical Activity of Cizutamig in Systemic Sclerosis
Brief Title: A Study of Cizutamig in Systemic Sclerosis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CND106-RUJN -1
Record Dates: First submitted 2025-08-25; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Systemic Sclerosis (SSc)
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A study of cizutamig in patients with Systemic Sclerosis (Ssc) (Experimental)
  Interventions: Drug: Biological: cizutamig

INTERVENTIONS:
Drug: Biological: cizutamig — Cizutamig will be dosed according to the protocol.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, PK, PD, immunogenicity, and preliminary clinical activity of cizutamig in patients with SSc.

DETAILED DESCRIPTION:
An Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Preliminary Clinical Activity of Cizutamig in Systemic Sclerosis

ELIGIBILITY:
ICriteria: Inclusion Criteria:

1. 18 to 75 years old at the time of signing the informed consent form (ICF)
2. Diagnosis of SSc according to the 2013 American College of Rheumatology (ACR)/ European Alliance of Associations for Rheumatology (EULAR) classification criteria
3. Diffuse cutaneous SSc according to the LeRoy criteria
4. Positive for at least 1 SSc-specific parameter as specified in the protocol
5. Disease duration of ≤ 7 years
6. mRSS ≥ 15
7. Inadequate response to therapies defined in the protocol.

Exclusion Criteria:

1. Inadequate clinical laboratory parameters at Screening
2. Receipt of or inability to discontinue any excluded therapies as specified in the protocol
3. Receipt of live vaccine within 4 weeks prior to Screening
4. Presence of any concomitant autoimmune disease other than the disease being studied
5. Receiving or anticipated to require total parenteral nutrition during the study
6. Active or history of intestinal pseudo-obstruction OR small intestinal bacteria overgrowth
7. Active or history of gastric antral vascular ectasia
8. Active digital ischemia with gangrene OR requiring antibiotics or amputation at Screening or during the study
9. Active or history of scleroderma renal crisis
10. History of progressive multifocal leukoencephalopathy
11. History of primary immunodeficiency or a hereditary deficiency of the complement system
12. Central nervous system (CNS) disease
13. Have presence of 1 or more significant concurrent medical conditions per investigator judgment
14. Have a diagnosis or history of malignant disease within 5 years prior to Screening
15. Inability to comply with contraception requirements as specified in the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-04 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) through end of study | 52weeks

IPD SHARING:
Plan to Share IPD: No